CLINICAL TRIAL: NCT03184844
Title: The Multi-center Clinical Trials of Thalidomide in TI
Brief Title: The Effective and Safety of Thalidomide in TI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiao-Lin Yin (Other)
Responsible Party: Sponsor-Investigator, Xiao-Lin Yin, Director, NO.3 Hospital of the People's Liberation Army, 303rd Hospital of the People's Liberation Army
Organization: 303rd Hospital of the People's Liberation Army (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 303 PLA
Record Dates: First submitted 2017-06-08; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Thalassemia
Keywords: Thalidomide TI
MeSH Terms: conditions — Thalassemia | interventions — Thalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- thalidomide thalassemia (Experimental): thalidomide:50mg/d p.o
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — thalidomide:50mg/d p.o at bedtime
  Other Names: fǎn yìng tíng

SUMMARY:
This is an exploratory experiment, aims to explore the effective and safety of thalidomide in the treatment of TI to improve the hemoglobin level, improve the quality of life, reduce blood transfusion, so as to avoid the adverse reactions caused by transfusion,60~100 patients will be enrolled.

DETAILED DESCRIPTION:
The project is a single arm research of thalidomide in TI,patients volunteered to participate in this trial and met the following inclusion criteria will be enrolled: age from 18~65, Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or less. Subjects should take thalidomide 50mg per day. During this time, hepatic and renal function, hematologic function, electrocardiogram and the adverse reactions were closely observed. According to the protocol, the blood routine, peripheral blood reticulocyte count, nucleated red blood cell count, hemoglobin electrophoresis and other indicators were evaluated in screening-period visit,1-month visit, 3-months visit , 6-months visit ,9-months visit, 12-months visit and 15-months visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting all of the following criteria will be considered for admission to the trial:

  * Diagnosis of NTDT;
  * Ages 18-65 years;
  * ECOG: 0~2 scores;
  * If not blood transfusion,the level of HB<90g/dl, or blood transfusion to maintain the HB;
  * Sign an informed consent agreeing to the clinical trial participation.

Exclusion Criteria:

* Patients presenting with any of the following criteria will not be included in the trial:

  * Patients received hydroxycarbamide, Yisui Shengxue Granule in three months;
  * Women during Pregnancy, breastfeeding or those of childbearing age who do not want to take contraceptive measures;
  * Patients had comorbidities like severe heart or lung diseases, liver dysfunction, cerebrovascular, cardiovascular, liver, kidney, tumor or other serious primary diseases;
  * Patients Allergic to the drug ingredients;
  * Patients with any Mental problem;
  * Patients had Participated in other drug clinical trials in the past 1 month;
  * Patients had a history of venous or arterial thrombosis;
  * In certain circumstances that the researchers determined it was not suitable for the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-02-02 (Estimated); Study Completion 2019-05-02 (Estimated)

PRIMARY OUTCOMES:
The Effective Rate of Patients | 24 months
  All participants will complete the treatment for 24 months, the hemoglobin value will be observed during the treatment,the value increased more than 20g/L defined as the marked effect,increased to 10~20g/L defined as effective, otherwise invalid.

SECONDARY OUTCOMES:
The Marked Improvement Rate of Patients | 24 months
  The highest hemoglobin value will be observed,the value increased more than 20g/L defined as the marked effect,increased to 10~20g/L defined as effective, otherwise invalid.

CONTACTS AND LOCATIONS:
Overall Officials: Yin X Lin, director, Study Director — NO.3 Hospital of the Chinese People's Liberation Army
Locations (1):
- NO.3 Hospital of the Chinese People's Liberation Army, Nanjing, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Twenty four months later after the last visit，summery report will be shared with other researchers through database

REFERENCES:
- [Derived] Ren Q, Zhou YL, Wang L, Chen YS, Ma YN, Li PP, Yin XL. Clinical trial on the effects of thalidomide on hemoglobin synthesis in patients with moderate thalassemia intermedia. Ann Hematol. 2018 Oct;97(10):1933-1939. doi: 10.1007/s00277-018-3395-5. Epub 2018 Jun 22. PMID 29931453